CLINICAL TRIAL: NCT01203150
Title: Exercise Treatment of Obesity-Related Secondary Conditions in Adults With Paraplegia
Brief Title: Effects of Exercise in People With Paraplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Mark S. Nash, Ph.D., FACSM, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TMP-MN-006
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supplement (Experimental): Participants randomized to the 'supplement' arm will consume a blended drink containing 48g of ionexchange, hydrolyzed vanilla-flavored whey protein (Whey to Go, Solgar Vitamin and Herb, Leonia, NJ; 3g CH2O, < 3g Total Fat). The drink will be given in split doses immediately before and after each training session, which represents a timing schedule that best stimulates muscle anabolism in persons undergoing exercise training.
  Interventions: Other: Exercise
- Placebo (Placebo Comparator): As ingestion of the protein supplement is critically influenced by time of administration, participants assigned to the 'placebo' study arm will consume the identical supplement and dose on days during which training is not performed. This strategy will allow the groups to be isocaloric and equal in protein supplementation.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — CRT will occur 3 times per week for 26 weeks. Each training session will last approximately 40-45 minutes and employ resistance training (weight lifting) and high-speed, low intensity endurance activities (arm cranking) with interposed periods of incomplete recovery (i.e., heart rate not falling to baseline).
  Other Names: Circuit Resistance Training (CRT)

SUMMARY:
This hypothesis-driven study will investigate effects of physical activity with or without a nutrient supplement known to increase body lean mass in adults with chronic paraplegia who have clusters of obesity and obesity-related secondary complications.

DETAILED DESCRIPTION:
Obesity and obesity-related secondary complications are pandemic health hazards that are highly prevalent among persons with spinal cord injuries (SCI). Accumulation of body fat disposes persons with SCI to accelerated endocrine and cardiovascular diseases, as well as pain, functional decline, and diminished health-related quality of life (HRQoL). While use of combined resistance and endurance exercise by persons without disability can remedy many of the problems associated with these disorders, their widespread use for persons with spinal cord injuries (SCI) must first satisfy scientific burdens of effectiveness.

The investigators have adopted the term "obesity-related secondary complications" to describe accumulation of body fat clustering with other secondary CVD risks, while recognizing that a threshold criterion for diagnosis of obesity in persons with SCI remains ill-defined. For purposes of this proposal, the "-related" part of the term confers physical deconditioning, hypertension, fasting dyslipidemia, post-prandial lipemia (PPL), and impaired insulin sensitivity, all of which have been reported in persons with SCI. Contextualized, any of these risks occurring independently or in clusters would be cause for immediate therapeutic lifestyle intervention (TLI), if not frank medical treatment. Given our early understanding of effective treatments for these risks, any improvement in their severity would be CVD risk-reducing and thus life-benefiting and function-preserving.

The investigators expect that the research findings will improve the understanding of risks for obesity and obesity-related secondary complications so that future interventions can be better targeted, identify an exercise intervention that can attend to current health risks, clarify whether nutrient supplementation improves risk-lessening benefits of exercise, identify exercise timing and intensities that best enhance fat utilization, and expand the understanding of the interrelated nature of risk factors after SCI.

ELIGIBILITY:
Inclusion Criteria:

* SCI resulting in paraplegia between T5 and L1
* injury for more than one year
* American Spinal Injury Association Impairment Scale (AIS) grade A-C injuries
* BMI ≥ 23 kg/m2 (defined by studies as the equivalent to the WHO criterion of 25 kg/m2 as 'overweight', and the point at which health risks begin to increase), plus any two or more of the following conditions on screening:

  1. prehypertension (BP ≥ 120/80 mmHg) by updated AHA and ADA criteria
  2. dyslipidemia (HDL-C ≥ 40 mg/dL or TG ≤ 150 mg/dL) by NCEP ATP III Guidelines,44 or
  3. impaired fasting glucose (≥ 100 mg/dL) by 2006 ADA criteria.

Exclusion Criteria:

* surgery within 6 months
* pressure ulcer within 3 months
* upper limb pain that limits exercise
* recurrent acute infection or illness requiring hospitalization or IV antibiotics
* pregnancy
* previous myocardial infarction or cardiac surgery
* 6 month history of glucose lowering and lipid-lowering drug therapy
* Type I or II diabetes (by WHO criteria)
* daily intake of vitamin supplements exceeding 100% RDA
* The following medications and drug therapies will disqualify subjects from participating: beta-adrenergic antagonists, maintenance alpha-blockers, Methyldopa, thiazide and loop diuretics, parasympatholytic agents, zinc, estrogen/hormone replacement therapy excluding oral contraceptives, insulin-sensitizing drugs, and maintenance use of aspirin and nonsteroidal anti-inflammatory drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Global cardiovascular disease risk score | 4 visits over 9 months
  Global cardiovacular disease risk will be generated by evaluating blood metabolism in the fasting and fed state for inflammatory disease markers including total cholesterol: high density lipoprotein ratio (TC: HDL ratio), post-prandial lipemia (PPL), whole body fat oxidation (WBFO), insulin resistance, and inflammatory mediators.

SECONDARY OUTCOMES:
Body composition | 4 visits over 9 months
  The percent of muscle and fat in each participants' body will be measured by dual x-ray absorptiometry (DEXA) scan.
Cardiovascular Endurance | 4 visits over 9 months
  Endurance will be measured using a calibrated upper arm ergometer. An initial exercise workload of 0 Watts at 60 revolutions per minute (RPM) for three minutes will be followed by three minute stages increasing in 20 Watt increments. Responses to exercise will be continuously monitored via open-circuit spirometry and 12-lead electrocardiography. Peak Work will be defined as volitional fatigue, inability to maintain targeted workload, or the point at which increasing workload fails to further increase VO2.
Muscular strength | 8 visits over 9 months
  Upper extremity dynamic strength testing will be performed on a Helms equalizer 1000 multi-station exerciser using the following maneuvers: overhead press, horizontal row, vertical butterfly, biceps curl, latissimus pull down (either to the chest or neck), and dips. The 1-repetition maximum (1-RM) will be calculated using the Mayhew regression equation.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nash, PhD, Principal Investigator — University of Miami Miller School of Medicine, The Miami Project to Cure Paralysis
Locations (1):
- The Miami Project to Cure Paralysis, Miami, Florida, United States